CLINICAL TRIAL: NCT00782184
Title: A Randomized, Double-Blind, Active-Controlled Study of Patients With Primary Hypercholesterolemia and High Cardiovascular Risk and Not Adequately Controlled With Atorvastatin: A Comparison of Switching to a Combination Tablet Ezetimibe/Simvastatin Versus Doubling the Baseline Dose of Atorvastatin
Brief Title: Ezetimibe/Simvastatin (10 mg/40 mg) vs. the Doubling of Atorvastatin in High Risk Participants (MK-0653A-134 AM1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-134; 2008_576
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Ezetimibe, Simvastatin Drug Combination; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ezetimibe/simvastatin 10/40 (Experimental): Participants received 20 mg open-label atorvastatin during a 5-week run-in period. Following this run-in period, ezetimibe/simvastatin 10/40 was administered once daily in tablet form during the 6-week double-blind treatment period
  Interventions: Drug: ezetimibe/simvastatin 10/40; Drug: atorvastatin 20 mg
- atorvastatin 40 mg (Active Comparator): Participants received 20 mg open-label atorvastatin during a 5-week run-in period. Following this run-in period, 40 mg atorvastatin was administered once daily in tablet form during the 6-week double-blind treatment period
  Interventions: Drug: atorvastatin 40 mg; Drug: atorvastatin 20 mg

INTERVENTIONS:
Drug: ezetimibe/simvastatin 10/40 — ezetimibe/simvastatin 10/40 tablet once daily for 6 weeks.
  Other Names: Vytorin
  Arms: ezetimibe/simvastatin 10/40
Drug: atorvastatin 40 mg — atorvastatin 40 mg tablet once daily for 6 weeks
  Other Names: Lipitor
  Arms: atorvastatin 40 mg
Drug: atorvastatin 20 mg — All participants will take atorvastatin 20 mg tablet once daily for the 5 week run-in period before randomization
  Other Names: Lipitor

SUMMARY:
Participants currently taking atorvastatin 20 mg will be switched to either atorvastatin 40 mg or ezetimibe/simvastatin 10 mg/40 mg (10/40). After 6 weeks of treatment, the percent reduction in low-density lipoprotein cholesterol (LDL-C) will be assessed and compared between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are either statin naive or on approved lipid lowering therapy for 6 weeks prior to study initiation
* Participant meets Adult Treatment Panel (ATP) III High Risk criteria

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Participant consumes more than 14 alcoholic beverages per week
* Participant has been treated with an investigational drug within the last 30 days
* Participant has congestive heart failure (New York Heart Association [NYHA] Type III or IV)
* Participant has had gastric bypass
* Participant is newly diagnosed with type 1 or 2 diabetes
* Participant is Human Immunodeficiency Virus (HIV) positive
* Participant has a history of drug or alcohol abuse within the last 5 years

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hing Ling PK, Civeira F, Dan AG, Hanson ME, Massaad R, De Tilleghem Cle B, Milardo C, Triscari J. Ezetimibe/simvastatin 10/40 mg versus atorvastatin 40 mg in high cardiovascular risk patients with primary hypercholesterolemia: a randomized, double-blind, active-controlled, multicenter study. Lipids Health Dis. 2012 Jan 31;11:18. doi: 10.1186/1476-511X-11-18. PMID 22293030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received 20 mg open-label atorvastatin during a 5-week run-in period.
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Started | 120 | 130
Completed | 116 | 125
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg | Total
Number analyzed (Participants) | 120 | 130 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.0) | 59.7 (8.4) | 59.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 65 | 122
  Male | 63 | 65 | 128

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Reaching LDL-C Target Goals of <70 mg/dL
Description: Target LDL-C level of < 70 mg/dL (1.81 mmol/L) at study endpoint after 6 weeks of treatment for the Full Analysis Set (FAS) population.
Time Frame: Treatment Week 6
Population: Participants in the Full Analysis Set (FAS) Population [all randomized participants with at least one dose of study treatment and baseline data] with baseline and post-baseline data available.
Measure: Number; unit: participants
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
participants | 34 | 6
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; COMPARISON BETWEEN GROUPS FOR NUMBER OF PARTICIPANTS REACHING LDL-C GOAL OF <70 MG/DL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.4, 95% CI 2-sided [3.4 to 21.0]

2. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein (LDL)-C
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: Participants in the Full Analysis Set (FAS) Population [all randomized participants with at least one dose of study treatment and baseline data] with percent change data available at week 6.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -26.81 (27.09) [-31.44 to -22.18] | -11.81 (22.85) [-16.40 to -7.22]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis (LDA) Model; Difference in Least Squares Means = -15.00, 95% CI 2-sided [-21.15 to -8.84]

3. Secondary Outcome: Number of Participants Reaching LDL-C Target Goal <77 mg/dL
Description: Target LDL-C level of < 77 mg/dL (2.00 mmol/L) at study endpoint after 6 weeks of treatment for the Full Analysis Set (FAS) population.
Time Frame: Treatment Week 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
participants | 45 | 11
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.7, 95% CI 2-sided [3.3 to 13.9]

4. Secondary Outcome: Number of Participants Reaching LDL-C Target Goal <100 mg/dL
Description: Target LDL-C level of < 100 mg/dL (2.59 mmol/L) at study endpoint after 6 weeks of treatment for the Full Analysis Set (FAS) population.
Time Frame: Treatment Week 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
participants | 81 | 52
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.5, 95% CI 2-sided [2.0 to 6.0]

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -15.97 [-19.17 to -12.76] | -7.73 [-10.91 to -4.55]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = -8.24, 95% CI 2-sided [-12.50 to -3.97]

6. Secondary Outcome: Percent Change From Baseline in Triglycerides
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -5.41 [-11.36 to 0.95] | -7.54 [-13.32 to -1.38]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.593, LDA Model; Difference in Least Squares Means = 2.13, 95% CI 2-sided [-5.67 to 9.93]

7. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein (HDL) Cholesterol
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | 5.37 [2.39 to 8.35] | 2.89 [-0.07 to 5.85]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.211, LDA Model; Difference in Least Squares Means = 2.48, 95% CI 2-sided [-1.41 to 6.37]

8. Secondary Outcome: Percent Change From Baseline in Non-HDL Cholesterol
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -22.50 [-26.78 to -18.22] | -10.88 [-15.13 to -6.64]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = -11.62, 95% CI 2-sided [-17.32 to -5.92]

9. Secondary Outcome: Percent Change From Baseline in LDL-Cholesterol/HDL-Cholesterol Ratio
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -28.77 [-33.78 to -23.76] | -12.66 [-17.63 to -7.69]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = -16.10, 95% CI 2-sided [-22.77 to -9.44]

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-Cholesterol Ratio
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -18.63 [-22.37 to -14.89] | -8.60 [-12.31 to -4.89]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = -10.02, 95% CI 2-sided [-14.96 to -5.08]

11. Secondary Outcome: Percent Change From Baseline in Non-HDL Cholesterol/HDL-Cholesterol Ratio
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -24.41 [-29.40 to -19.43] | -11.20 [-16.15 to -6.25]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = -13.21, 95% CI 2-sided [-19.83 to -6.59]

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -17.23 [-20.84 to -13.62] | -9.53 [-13.12 to -5.95]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.002, LDA Model; Difference in Least Squares Means = -7.69, 95% CI 2-sided [-12.50 to -2.88]

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | 2.56 [0.36 to 4.77] | -2.69 [-4.88 to -0.50]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = 5.25, 95% CI 2-sided [2.44 to 8.06]

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/A-1 Ratio
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -18.59 [-22.70 to -14.48] | -5.67 [-9.76 to -1.59]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, LDA Model; Difference in Least Squares Means = -12.91, 95% CI 2-sided [-18.31 to -7.52]

15. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-Reactive Protein (Hs-CRP)
Time Frame: Baseline (Treatment Day 1), Treatment Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg
Number analyzed (Participants) | 117 | 126
percent change from baseline | -6.18 [-20.49 to 10.70] | -8.86 [-22.67 to 7.41]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.785, LDA Model; Difference in Least Squares Means = 2.68, 95% CI 2-sided [-16.50 to 21.86]

ADVERSE EVENTS:
Groups:
- Placebo: One participant received 20 mg open-label atorvastatin during a 5-week run-in period. Following this run-in period, the participant was randomized to the ezetimbe/simvastatin group, but took only pills from the bottle containing placebo to atorvastatin during the 6-week double-blind treatment period.
Arm/Group | Ezetimibe/Simvastatin 10/40 | Atorvastatin 40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/119 | 1/130 | 0/1
Other Adverse Events (participants affected / at risk) | 0/119 | 2/130 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin 10/40 (N=119) | Atorvastatin 40 mg (N=130) | Placebo (N=1)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin 10/40 (N=119) | Atorvastatin 40 mg (N=130) | Placebo (N=1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.